CLINICAL TRIAL: NCT05833789
Title: Visualization of the Colon Through Use of the Magnetic Flexible Endoscope (MFE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Keith Obstein, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MFE_222293; 5R01EB018992-07 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-04-27 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Colon; Robotic; Magnetic; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Colonoscopy for colorectal cancer screening (Experimental): All patients in this group will have their colonoscopy for colorectal cancer screening completed with a legacy colonoscope followed by colonoscopy with the Magnetic Flexible Endoscope (MFE).
  Interventions: Device: Magnetic Flexible Endoscope (MFE)

INTERVENTIONS:
Device: Magnetic Flexible Endoscope (MFE) — After colonoscopy has been completed with the legacy colonoscope, the MFE will be introduced into the colon and traverse from the rectum to the cecum.

SUMMARY:
In this study, the investigators will evaluate the ability of the Magnetic Flexible Endoscope (MFE) to travel through the human colon. The MFE is a device made of ultra-flexible tubing that contains a camera, light, and magnet at the tip. The tip of the tube is about the size of a penny. The magnet inside the tip allows the MFE to be moved through the colon by a second magnet attached to a robotic arm that is outside the body. The objective of this feasibility study is to determine navigation of the colon and tolerability of the Magnetic Flexible Endoscope (MFE) traveling in the human colon.

DETAILED DESCRIPTION:
The clinical practice at Vanderbilt University Medical Center (VUMC) is to perform the screening colonoscopic exam while the patient is sedated (Monitored Anesthesia Care administered by the VUMC out-of-OR Anesthesia team) with a legacy colonoscope (Olympus CF/PCF-H190L; Olympus America, Center Valley, PA, USA) to evaluate the patient's colon (via the rectum passed trans-anally with the intent of reaching the cecum). After the screening examination with the legacy colonoscope has been completed and the legacy colonoscope is removed from the patient, the sedation for the patient is stopped as per the standard of care. The patient will be monitored as per VUMC standard of care post-sedation monitoring protocol in the procedure room (post-sedation recovery phase). While the patient is in the post-sedation recovery phase in the procedure room, the MFE will be inserted trans-anally into the rectum and traverse the colon with the intent on reaching the cecum. No additional sedation is administered. After the cecum is visualized, the MFE will be removed from the patient. The patient will continue to be monitored as per VUMC standard of care post-procedure monitoring protocol in the procedure room. Once VUMC standard of care discharge parameters have been met, the patient will be discharged from the procedure area/VUMC as per standard of care. The investigators plan to enroll 5 healthy patients who are already scheduled to undergo their standard of care colonoscopic exam for age-appropriate colorectal cancer screening. The endpoints of the study are navigation of the colon, mucosal visibility, tolerability of the MFE traveling in the human colon, and endoscopist assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 70 years of age.
2. Able to provide written informed consent.
3. ASA class < 3
4. No significant medical problems
5. Abdominal circumference < 96 cm

Exclusion Criteria:

1. Patients who do not meet inclusion criteria
2. Patients who are unable or unwilling to provide informed consent
3. Magnetic implants and wearable devices (such as insulin pumps)
4. Patients who are pregnant. As part of routine pre-operative care, all patients with uterus who are of childbearing potential will undergo either urine or blood pregnancy testing
5. Cancer positive subjects or any patients currently undergoing any treatment or therapy to treat, cure, or mitigate cancer
6. Symptoms consistent with coronavirus (COVID-19) --- pyrexia, new persistent cough or anosmia --- or a positive coronavirus (COVID-19) PCR swab result
7. Previous failed colonoscopy
8. Colonic resection
9. Severe diverticulosis
10. Known or suspected colonic stricture
11. Previous radiation therapy to the abdomen or pelvis
12. Any active inflammatory bowel condition (e.g. active IBD or diverticulitis)
13. Known or suspected bowel obstruction
14. Presence of ascites
15. Participants taking anticoagulant medications or antiplatelet therapy (excluding aspirin) within the last 7 days
16. Known coagulation disorder (INR ≥ 1.5 or platelets < 150 x 10^9)
17. Known to have phenylketonuria or G6PD deficiency
18. Abdominal surgery within the last 6 months
19. Drug or alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith L Obstein, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Obstein KL, Landewee CA, Martin J, Calo S, Norton J, Wai Kow J, Scaglioni B, Valdastri P. The Magnetic Flexible Endoscope: Phase 1 First-in-Human Clinical Trial. Am J Gastroenterol. 2025 Jun 10:10.14309/ajg.0000000000003584. doi: 10.14309/ajg.0000000000003584. Online ahead of print. PMID 40493042

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colonoscopy for Colorectal Cancer Screening
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colonoscopy for Colorectal Cancer Screening
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: MFE Navigation to the Cecum From the Rectum in Less Than 40 Minutes
Description: Number of participants with successful MFE navigation to the cecum from the rectum of the colon in less than 40 minutes
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Colonoscopy for Colorectal Cancer Screening
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: MFE Tolerability by Post-procedure Interview
Description: Number of reported non-tolerability events, including events associated with the product's administration affecting the ability or desire of the patient to adhere to the intensity of therapy. Tolerability was assessed through qualitative interview post procedure.
Time Frame: Day 1
Measure: Number; unit: events
Arm/Group | Colonoscopy for Colorectal Cancer Screening
Number analyzed (Participants) | 5
events | 0

3. Secondary Outcome: Endoscopist Experience by NASA Task Load Index (TLX)
Description: The NASA Task Load Index (TLX) is a validated assessment instrument (Ames Research Center, Moffett Field, CA, USA) to assess perceived workload based on a multidimensional construct of six sub-scales: mental demand, physical demand, temporal demand, performance, effort, and frustration level. The sub-scales range from 0 (very low) to 100 (very high); the exception is the sub-scale of performance, where 0 is perfect and 100 is failure.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Colonoscopy for Colorectal Cancer Screening
Number analyzed (Participants) | 5
score on a scale
  Mental | 31 [28 to 33]
  Physical | 44 [29 to 47]
  Temporal | 28 [25 to 31]
  Performance | 47 [46 to 47]
  Effort | 36 [29 to 45]
  Frustration | 40 [32 to 45]

4. Secondary Outcome: Colon Mucosal Visibility
Description: Colon mucosal visibility scale is an operator assessed cumulative score utilizing the colon visualization index which has a score range of 0-4, where 0 is poor and 4 is excellent.
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Colonoscopy for Colorectal Cancer Screening
Number analyzed (Participants) | 5
score on a scale | 3 [2.8 to 3]

ADVERSE EVENTS:
Time Frame: Day 1
Arm/Group | Colonoscopy for Colorectal Cancer Screening
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05833789/Prot_001.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT05833789/SAP_002.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT05833789/ICF_000.pdf